CLINICAL TRIAL: NCT00183742
Title: Phase I Trial of Liposomal Doxorubicin (Doxil) and Weekly Docetaxel (Taxotere)
Brief Title: Trial of Liposomal Doxorubicin (Doxil) and Weekly Docetaxel (Taxotere)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0C-00-6
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Cancer; Carcinoma
Keywords: Phase 1; Phase I; Phase one; Solid tumor
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — liposomal doxorubicin; Docetaxel

INTERVENTIONS:
Drug: liposomal doxorubicin and docetaxel

SUMMARY:
This study is for patients with advanced cancer that has failed treatment with conventional therapy or for which no standard treatment exists. The purpose of this study is to determine the highest dose that can be given of 2 chemotherapy drugs, docetaxel (also called Taxotere) and liposomal doxorubicin (also called Doxil), when given together and to determine the side effects of this combination. Both Taxotere and Doxil are chemotherapy drugs that can decrease the size of several different tumors. Taxotere is approved by the Food and Drug Administration (FDA) for the treatment of breast and lung cancers, and Doxil is approved for the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of advanced or recurrent solid tumor which has failed prior therapy, or for which no effective therapy is available.
* Ovarian cancer patients (or primary peritoneal carcinoma) whose only manifestation of disease is an elevated cancer antigen (CA) 125 of > 100 are eligible.
* SWOG performance status 0-2.
* Absolute granulocyte count (AGC) greater than or equal to 1.5; platelets greater than or equal to 100,000.
* Total bilirubin less than or equal to the upper limit of normal (ULN).
* Transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is <= ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are <= ULN. However, patients who have both transaminase elevation > 1.5 x ULN and alkaline phosphatase > 2.5 x ULN are not eligible for this study (due to decreased clearance of docetaxel and increased risk of toxicity).
* Age greater than or equal to 18 years.
* Fully recovered from acute toxicities from chemotherapy, radiation, or surgery.
* Negative serum pregnancy test, if patient is female, still fertile, and sexually active.

Exclusion Criteria:

* Prior treatment with Doxil or weekly docetaxel. Prior docetaxel administered every 3 weeks is allowed.
* Evidence of moderate peripheral neuropathy greater than or equal to grade 2.
* Medical, social, or psychological factors interfering with compliance.
* Known history of cardiac disease (congestive heart failure, coronary artery disease) that would preclude treatment with Doxil in the opinion of the investigator.
* Cardiac ejection fraction < 50%
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2000-12; Primary Completion 2005-10 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of liposomal doxorubicin (Doxil) administered every 4 weeks or every 2 weeks in combination with docetaxel (Taxotere) administered on a weekly schedule
To establish the toxicity profile of this combination

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C./Norris Comprehensive Cancer Center
Locations (1):
- U.S.C./Norris Comprehensive Cancer Center, Los Angeles, California, United States